CLINICAL TRIAL: NCT00906113
Title: Phase 1-2 Study of Injection of Melphalan Into the Ophthalmic Artery in Children With Retinoblastoma
Brief Title: Intra-arterial Chemotherapy for Children With Retinoblastoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Michael Weintraub, DIrector, Pediatric Hematology Oncology, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0058-09-HMO
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intra-arterial melphalan (Experimental): The patients will be treated by injection of chemotherapy (melphalan) into the ophthalmic artery of an eye affected by retinoblastoma
  Interventions: Drug: Intra-arterial injection of melphalan; Drug: Injection of melphalan into the ophthalmic artery

INTERVENTIONS:
Drug: Intra-arterial injection of melphalan — Injection of 5 milligrams of melphalan into the ophthalmic artery once every 3 weeks for a total of 6 courses
Drug: Injection of melphalan into the ophthalmic artery — Injection of 5 milligrams of melphalan into the ophthalmic artery in an eye affected by retinoblastoma

SUMMARY:
Retinoblastoma is a cancer of the eye that occurs exclusively in children. The treatment for retinoblastoma may include surgery, chemotherapy, radiation and local treatments to the eye such as freezing (cryotherapy) and local radiation (brachytherapy). In some cases, a child with retinoblastoma will have active cancer in a single remaining eye with useful vision. In such cases, it is sometimes necessary to remove this eye. In such cases, the injection of chemotherapy directly into the artery that supplies the eye and the tumor may lead to regression of the tumor without the need to remove the eye.

This form of treatment was pioneered by a group in New York (Abramson et al). In this study the investigators will assess the efficacy and safety of the technique in a group of children with retinoblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Children with retinoblastoma in a single remaining eye with useful vision

Exclusion Criteria:

* None

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2011-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Salvage of eye and vision | Three years from intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes